CLINICAL TRIAL: NCT05415800
Title: Facilitation of Cancer Prevention and Screening Guideline Implementation: Pilot Study
Brief Title: Quality Improvement Pilot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela Hull, Associate Professor, University of Kentucky
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 77178; 3P30CA177558-08S3 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): Intervention
  Interventions: Behavioral: Quality Improvement Practice Facilitation Intervention

INTERVENTIONS:
Behavioral: Quality Improvement Practice Facilitation Intervention — The practice facilitation intervention (implementation strategy package) consists of QI projects designed for primary care providers with external practice facilitation and technical support provided by a QI Coach and Data Coach on our team.
  The QI projects focus on the implementation of cancer prevention and early detection guidelines in primary care settings, specifically one QI project for each of the following clinical guidelines: colorectal cancer screening, lung cancer screening, and tobacco treatment. The study participants are the healthcare providers and staff, not the patients, since the goal of the practice facilitation intervention (implementation strategy package) is to improve the implementation of existing standard of care.

SUMMARY:
The overall goal of this study is to develop and pilot test the use of practice facilitation as an intervention for healthcare providers and staff, with the goal of improving the implementation of cancer prevention and screening guidelines in primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Normal Volunteers

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal Cancer: Screening Rate (Patient Population) | 6 months
  Percent of patients age 50-75 who completed appropriate screening for colorectal cancer.
Lung Cancer: Screening Rate (Patient Population) | 6 months
  Percent of eligible patients with shared decision-making visit AND completed baseline LDCT scan.
Tobacco: Treatment Rate (Patient Population) | 6 months
  Percent of patients identified as tobacco user who received tobacco cessation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Hull, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States